CLINICAL TRIAL: NCT01970280
Title: Low Molecular Weight Heparin in Prevention of Recurrent Arteriovenous Graft Thrombosis in Chronic Hemodialysis Patients.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr. Sidney Ben Chetrit (Other)
Responsible Party: Sponsor-Investigator, Dr. Sidney Ben Chetrit, MD, Meir Hospital, Kfar Saba, Israel
Organization: Meir Hospital, Kfar Saba, Israel (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0146-13-MMC; 0146-13-MMC (Other: Meir Medical Center, Nephrology and hypertension department, Kfar Sava, Israel)
Record Dates: First submitted 2013-10-22; First posted 2013-10-28 (Estimated); Last update posted 2013-10-28 (Estimated); Status verified 2013-10

CONDITIONS: Hemodialysis Patients
MeSH Terms: interventions — Enoxaparin

ARMS (2):
- Enoxaparin (Active Comparator): Following a first AV graft thrombosis and successful thrombolysis with angioplasty, patients on chronic hemodialysis will be randomized to s.c Enoxaparin (Clexane) 0.5 mg/1kg of body weight per day or control group (not on Clexane).
  Interventions: Drug: Enoxaparin
- Observation (No Intervention)

INTERVENTIONS:
Drug: Enoxaparin
  Arms: Enoxaparin

SUMMARY:
The aim of the study is to evaluate the effect of Enoxaparin (LMWH) on the incidence of AV graft thromboses in patients on chronic hemodialysis.

Primary efficacy end point of the study: to compare the time of onset of a new thrombotic event after successful angiography of the AV graft.

Pprimary safety outcome of the study: frequency of hemorrhage. Design and methods: Following a first AV graft thrombosis and successful thrombolysis with angioplasty, patients on chronic hemodialysis will be randomized to s.c Enoxaparin (Clexane) 0.5 mg/1kg of body weight per day or control group (not on Clexane). Patients will be followed for a year or till next AV graft thrombotic occlusion, if it occurs before. In both groups we will compare time periods in months between first and recurrent thrombotic events of AVG by evaluation the difference between two sample means. Also interim analysis of AV grafts patency between the two groups will be evaluated at different time points: three, six and twelve months after randomization. Patients in both groups will receive unfractionated heparin during dialysis session to prevent thrombosis of extracorporeal circulation. Patients from Enoxaparin group will receive a half dose (500 units/hour) to prevent possible risk of bleeding during the session. Before randomization all patients will be evaluated for hypercoagulability state which will include: Factor V Laden deficiency, Anti phospholipid antibodies (APLA), Antithrombin III deficiency and Protein C/S deficiency.

ELIGIBILITY:
Inclusion Criteria:

* hemodialysis patients ≥ 18 years of age after occurrence of AVG thrombosis and successful thrombolysis/thrombectomy with angioplasty.

Exclusion Criteria:

1. Known allergy to enoxaparin
2. Persistent systolic blood pressure 180 or more and/or persistent diastolic blood pressure 100 or more
3. Chronic Warfarin treatment
4. Double antiagregant treatment (aspirin plus clopidogrel)
5. Platelets count below 80000/µl
6. Known HIT (Heparin Induced Thrombocytopenia)
7. Recent bleeding (<2 weeks)
8. Recent stroke (<4 weeks)
9. Reduced mental status and inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-11 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
To compare the time of onset of a new thrombotic event after successful angiography of the AV graft. | 1 y

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Department of Nephrology and Hypertension, Meir Medical Center, Kfar Saba
  - Helsinki committee, Kfar Saba